CLINICAL TRIAL: NCT00412698
Title: A European Randomized, Parallel Group, Two-arm Placebo-controlled, Double-blind Multicenter Study of Rimonabant 20mg Once Daily in the Treatment of Abdominally Obese Patients With Dyslipidemia With or Without Other Comorbidities
Brief Title: European Trial About Effect of RimoNabant on Abdominal Obese Patients With dysLipidemia
Acronym: ETERNAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision has been taken in light of recent demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIMON_R_00962; EUDRACT # : 2006-001715-30
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Obesity; Dyslipidemias
MeSH Terms: conditions — Obesity; Dyslipidemias | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rimonabant
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rimonabant — Administration of one tablet containing 20 mg of active rimonabantonce daily in the morning.
  White film-coated tablets, for oral administration containing 20 mg of active rimonabant
  Arms: 1
Drug: Placebo — Administration of one rimonabant placebo tablet once daily in the morning. Undistinguishable placebo tablets.
  Arms: 2

SUMMARY:
Primary :

To determine the effect of Rimonabant 20 mg on changes in, HDL-Cholesterol (HDL-C), triglyceride levels over a period of 12 months when prescribed with a mild hypocaloric diet in abdominally obese patients with dyslipidemia with or without other associated comorbidities.

Main Secondary :

To determine the effect of 12 months Rimonabant treatment versus placebo on changes in waist circumference (WC), body weight, glycemic and lipid parameters.

To assess the safety of 12 months Rimonabant treatment versus placebo in these patients.

In selected sites, a sub study will be conducted to determine the effect of 12 months of Rimonabant on additional lipoprotein and inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27 kg/m² and < 40 kg/m²,
* Waist Circumference > 88 cm in women; > 102 cm in men,
* HDL cholesterol < 40 mg/dL (1.03 mmol/L) for men; < 50 mg/dL (1.29 mmol/L) for women, and/or Triglycerides ≥ 150 mg/dL (1.69 mmol/L),
* LDL cholesterol up to 155 mg/dl (4.00 mmol/L) including patients on a stable dose of statins and/or Ezetimibe therapy for at least 8 weeks prior to screening

Concomitant medications:

* Current treatment with statins and/or ezetimibe and/or antihypertensive therapy must be at fixed and stable dose for at least 8 weeks prior to screening visit,
* Patients, who are willing and in the opinion of the Investigator safely assumed to remain on stable and fixed doses of antihypertensive, and/or statins and/or ezetimibe without adding additional medications or changing current treatment for the duration of the trial.

Exclusion Criteria:

* Pregnant or breast-feeding women, or women planning to become pregnant or breastfeed (excluded by pregnancy test),
* Absence of medically approved contraceptive methods for female of childbearing potential,
* History of very low-calorie diet within 3 months prior to screening visit (lower than 1200 Kcal/day),
* Weight change > 5 kg within 3 months prior to screening visit,
* History of surgical procedures for weight loss (e.g., stomach stapling, bypass),
* History of bulimia or anorexia nervosa as per DSM-IV criteria
* Presence of any clinically significant endocrine disease according to the investigator, in particular known abnormal TSH and free T4 blood level (Patients treated with thyroid replacement therapy must be on fixed and stable dose for at least 3 months prior to screening and must be in euthyroïd status),
* Established type 1 or 2 diabetes treated, or with at least 2 measures of fasting blood glucose ≥ 126 mg/dl,
* Triglyceride level > 400 mg/dL (4.52 mmol/L),
* Systolic blood pressure > 160 mm Hg or diastolic blood pressure >100 mmHg at screening visit,
* Known severe renal dysfunction (creatinine clearance < 30 ml/min) or nephrotic syndrome or urinalysis (performed at screening by dipstick) showing 2+ or more protein,
* Known severe hepatic impairment or AST and/or ALT > 3 times the upper limit of normal at screening,
* Presence of any condition (medical, including clinically significant abnormal laboratory tests, psychological, social or geographical) actual or anticipated that the investigator feels would compromise the patient's safety or limit his/her successful participation to the study. In particular :

  * Cardiac abnormalities: cardiac failure status NYHA III or IV, relevant acute abnormal finding seen on ECG at screening or within 6 months before screening,
  * Any current malignancy or any cancer within the past five years (except adequately treated basal cell skin cancer or cervix carcinoma in situ),
  * Significant haematology abnormalities (haemoglobin < 100 g/L and/or neutrophils < 1.5 G/L and/or platelets < 100 G/L),
  * Acute psychiatric disorders, or mental condition which could interfere with the patient's compliance or safe participation in the study,
  * Patient treated for epilepsy
* Ongoing major depressive illness,
* Uncontrolled psychiatric illness,
* History of alcohol or other substance abuse,
* Hypersensitivity /intolerance to the active substance or to any of the excipients such as lactose,

Concomitant medications prior to study entry::

* Administration of any investigational treatment (drug or device) within 30 days prior to screening,
* Previous participation in a Rimonabant study or previous administration of Rimonabant,
* Administration of any of the following within 3 months prior to screening visit:

  * anti obesity drugs (eg, sibutramine, orlistat),
  * other drugs for weight reduction (phentermine, amphetamines),
  * herbal preparations for weight reduction,
  * nicotinic acid, fibrates or bile acid sequestrants,
  * Prolonged use (more than one week) of systemic corticosteroids, neuroleptics,
  * Omega-3 fatty acid approved medication
* Ongoing antidepressive treatment (including bupropion)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in HDL-C and triglyceride levels | From baseline to end of treatment

SECONDARY OUTCOMES:
Waist circumference and body weight | At each visit
Glycemic parameters : FPG, fasting insulinemia, HbA1c, | Prior to baseline, month 3, month 6 and month 12.
Lipid parameters : Total Cholesterol, HDL-C, LDL-C, triglyceride levels | Prior to baseline, month 3, month 6 and month 12.
Inflammatory parameter : Hs-CRP | Prior to baseline, month 3, month 6 and month 12.
Quality of life : IWQOL questionnaire completed | At baseline, month 3, month 6, month 9 and month 12.
Incidence of adverse events in each group, including neuro-psychiatric adverse events | Prior to baseline, month 3, month 6 and month 12.
Standard laboratory assessments | Prior to baseline and month 12
In selected sites, a sub study will be conducted in which additional Lipid parameters will be measured: HDL subfractions, Apo A1, Apo A2, Apo B and Apo C3, Lp A1, LpA1/A2, Lp(a), Oxidized-LDL and LDL size | Prior to baseline and at month 12
In selected sites, a sub study will be conducted in which additional Inflammatory parameters will be measured: Adiponectin-High Molecular Weight, Intracellular adhesion molecule 1(ICAM-I) and TNFalpha. | Prior to baseline and at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Stockholm, Sweden
- Sanofi-Aventis Administrative Office, Meyrin, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom